CLINICAL TRIAL: NCT05563610
Title: Oral Penicillin Challenge and Allergy De-labeling in the Phoenix Children's Hospital Emergency Department
Brief Title: Oral Penicillin Challenge and Allergy De-labeling in Children
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit sufficient number of subjects in the setting
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Principal Investigator, Diane E. Hindman, MD, Attending Physician, Phoenix Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-22-154
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Penicillin Allergy
Keywords: penicillin; anaphylaxis; allergy; oral challenge; amoxicillin; pediatric; emergency department
MeSH Terms: conditions — Anaphylaxis; Hypersensitivity; Emergencies | interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Challenge (Experimental): Patients will be screened for high vs. low risk of penicillin allergy. Low risk patients will be randomized to oral amoxicillin 500 mg challenge.
  Interventions: Drug: Amoxicillin 500mg
- No Oral Challenge (No Intervention): Patients will be screened for high vs. low risk of penicillin allergy. Low risk patients will be randomized to no oral amoxicillin 500 mg challenge..

INTERVENTIONS:
Drug: Amoxicillin 500mg — Patients screened to be low risk of penicillin allergy will be randomized to receive amoxicillin dose or not
  Other Names: Oral Challenge
  Arms: Oral Challenge

SUMMARY:
The primary purpose of this study is to investigate the portion of penicillin allergy labels that are not true allergies using oral amoxicillin challenges among pediatric patients. The secondary purpose is to evaluate the safety and feasibility of administering oral penicillin allergy challenges in the Pediatric Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in the pediatric emergency department who are 2-17 yo and labeled as penicillin-allergic (including amoxicillin or other penicillin allergies)
2. Patients at low risk of anaphylaxis as determined by the study questionnaire
3. Patients who would normally be prescribed amoxicillin, amoxicillin-clavulanate or another penicillin for their current bacterial infection, including otitis media, Group A Streptococcal pharyngitis, pneumonia. sinusitis, dog and cat bite wounds, regimens for Helicobacter pylori eradication, or other acute infections deemed susceptible.
4. Patients who are interested in participating
5. Patients who have an acceptable surrogate to give consent on the subject's behalf
6. Patients whose surrogate (parent/caregiver) speaks English or Spanish

Exclusion Criteria:

1. Patients who are uninterested in participating, or their parents/caregivers are not interested in having them participate
2. Patients who have multiple drug allergies

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Participants are eligible based on their self-representation of gender identity.
Enrollment: 31 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
True Penicillin Allergies | 24 hours after amoxicillin oral challenge
  Percentage of study patients presenting to the pediatric ED who received the amoxicillin oral challenge who demonstrated a true IgE-mediated allergic reaction

SECONDARY OUTCOMES:
Amoxicillin Oral Challenge Safety - High-Risk Reactions | 24 hours after amoxicillin oral challenge
  Percentage of high-risk penicillin allergic reactions
Amoxicillin Oral Challenge Safety - Admissions | 24 hours after amoxicillin oral challenge
  Percentage of admissions from the pediatric ED in patients experiencing high-risk penicillin allergic reactions
Amoxicillin Oral Challenge Safety - Re-admissions | 24 hours after amoxicillin oral challenge
  Percentage of re-admissions from home after discharge from the pediatric ED in patients experiencing high-risk penicillin allergic reactions
Amoxicillin Oral Challenge Safety - Deaths | 24 hours after amoxicillin oral challenge
  Percentage of deaths in patients experiencing high-risk penicillin allergic reactions
Amoxicillin Oral Challenge Feasibility | 24 hours after amoxicillin oral challenge
  Average hospital length of stay in the pediatric ED for patients receiving the amoxicillin oral challenge relative to the non-treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Diane E Hindman, MD PharmD, Principal Investigator — Emergency Department Attending Physician
Locations (1):
- Phoenix Children's, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers at this time.